CLINICAL TRIAL: NCT04528108
Title: Efficacy Evaluation of Kidney-tonifying and Tune up Chong-Ren Hemostasis Chinese Medicine Periodic Therapy for Dysfunctional Uterine Bleeding During Adolescence With Yin Deficiency and Blood Heat Syndrome: a Randomized Controlled Study
Brief Title: Chinese Medicine Periodic Therapy for Dysfunctional Uterine Bleeding During Adolescence With Yin Deficiency and Blood Heat Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19401931000
Record Dates: First submitted 2020-08-22; First posted 2020-08-27 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-04

CONDITIONS: Dysfunctional Uterine Bleeding
MeSH Terms: conditions — Metrorrhagia

STUDY DESIGN:
Intervention Model Description: In our research, 160 children are randomly divided into a Chinese medication periodic therapy group and a Gong Xue Ning control group, and they receive different treatment for 3 month.
Who Masked: Participant, Outcomes Assessor
Masking Description: In our research, participants and outcome assessor are are prevented from having knowledge of the interventions assigned to individual participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ZYZQ Group (Experimental): ZYZQ group is the experimental group which is treated with kidney-tonifying and tune up Chong-Ren hemostasis Chinese medicine for 3 months.
  Interventions: Drug: Kidney-tonifying and tune up Chong-Ren hemostasis Chinese medicine
- GXN Group (Active Comparator): GXN group is the active Comparator group which is treated with Gong Xue Ning capsules for 3 months
  Interventions: Drug: Gong Xue Ning capsules

INTERVENTIONS:
Drug: Kidney-tonifying and tune up Chong-Ren hemostasis Chinese medicine — Participants of Chinese medicine periodic therapy group will be treated with kidney-tonifying and tune up Chong-Ren hemostasis Chinese medicine periodic therapy. During bleeding period, use kidney-tonifying, heat-clearing and consolidating channel for hemostasis Chinese medicine to stop bleeding. The kidney-tonifying hemostasis prescription is made up of Nvzhenzi, Hanliancao, Tusizi, Xianhecao, Cebaiyetan, Danpi, Zhimu, etc. When the bleeding stops, use the kidney-tonifying, essence-strengthening and blood-activating, menstruation-regulating Chinese medicine to regulate menstruation. The kidney-tonifying and menstruation-regulating prescription is made up of Shengshudi, Zhimu, Tusizi, Fupenzi, Bajirou, Danggui, Danpi, etc. The drugs are granules for taking after infusion once a day. Participants receive this treatment for 3 months.
  Arms: ZYZQ Group
Drug: Gong Xue Ning capsules — Participants of Gong Xue Ning capsules group children will be treated with Gong Xue Ning capsules, 2 capsules 3 times a day during the bleeding period. When the bleeding stops, patients will be treated with Zhi Bai Dihuang pills,8 pills 3 times a day. Participants receive this treatment for 3 months.
  Arms: GXN Group

SUMMARY:
The purpose of this study is to conduct a randomized, single blind, controlled intervention trial to observe the therapeutic effect of kidney-tonifying and tune up Chong-Ren hemostasis Chinese medicine periodic therapy for dysfunctional uterine bleeding based on objective Chinese and western medicine evaluation standard.

DETAILED DESCRIPTION:
Dysfunctional uterine bleeding during adolescence is the most common menstrual disorders during adolescence, and the age of children suffering from it tended to be lower. It's urgent to explore effective ways to alleviate the pain caused by dysfunctional uterine bleeding.

In our research, 160 children are randomly divided into a Chinese medication periodic therapy group (80 cases) and a Gong Xue Ning control group (80 cases). Paticipants in Chinese medication periodic therapy group are treated with kidney-tonifying and tune up Chong-Ren hemostasis Chinese medicine for 3 months, whereas the Gong Xue Ning control group received Gong Xue Ning capsules for 3 months. We compare the effect of the two therapies about hemostasis and menstruation regulation, and the change of the thickness of endometrium, sex hormones, Kisspeptin, and PAI-1 in blood before and after the treatment, in order to make clear the efficacy and the mechanism of the Chinese medicine periodic therapy.

ELIGIBILITY:
Inclusion Criteria:

* satisfy the diagnostic criteria in the textbook<Obstetrics and Gynecology> with dysfunctional uterine bleeding
* age between 10-18 years
* course of the disease is 2 months or more.

Exclusion Criteria:

* have uterine bleeding on account of systemic diseases or organic diseases in reproductive system, such as blood diseases, thyroid diseases, hepatic diseases, etc.
* HB<80g/L
* have mental disorders
* allergic to many kinds of drugs

Ages: 10 Years to 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — This condition of the study is dysfunctional uterine bleeding, so we can only include female participants in our study.
Enrollment: 160 (Actual)
Dates: Start 2020-09-02 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Restoration of menstruation cycle(binomial) | the end of the third months
  Restoration of menstruation cycle is a binomial variable. Through clinical follow-up and menstrual diary, we record participants' menstrual period at month 3 of the treatment to confirm the restoration of menstruation, and we regard the menstrual cycle that is within 25-35 days as a normal cycle. Then normal cycles are defined as 1, and the rest are defined as 0.

SECONDARY OUTCOMES:
Menstrual hemostatic time | during procedure (about 3 months)
  We give every patient a menstrual diary to record the length of menstrual bleeding every month in order to confirm the hemostatic time.
Menstrual blood volume | during procedure (about 3 months)
  Menstrual blood volume is a repeated measurement variable. We give every participant a pictorial blood loss assessment chart (PBAC) to measure the menstrual blood volume. They fill in the chart every day during menstrual period according to the degree to which each item of sanitary protection was soiled with blood, thus we can calculate a score and speculate the menstrual blood volume based on that.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No